CLINICAL TRIAL: NCT01721499
Title: Decreasing Stress and Improving Self-control With "Stress in Control" (Sync) Training
Acronym: Sync
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Rajita Sinha, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0809004271
Record Dates: First submitted 2012-03-08; First posted 2012-11-05 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Stress; Obesity; Overeating
Keywords: Stress; obesity; overeating
MeSH Terms: conditions — Obesity; Hyperphagia | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness intervention (Experimental): The mindfulness intervention consists of weekly group format mindfulness instruction and skills development, weekly individual therapy sessions, and 6 nutritional sessions.
  The control group receives 6 nutritional sessions only.
  Interventions: Behavioral: Nutritional Counseling; Behavioral: Mindfulness Intervention
- Nutrition Control Group (Active Comparator): The control group receives 6 nutritional counseling sessions.
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Behavioral: Nutritional Counseling — weekly group and individual skills training to improve self control and decrease stress.
Behavioral: Mindfulness Intervention
  Arms: Mindfulness intervention

SUMMARY:
This is a study of treatment approaches aimed to improve self-control and decrease stress and unhealthy/maladaptive behaviors such as drinking, overeating, and smoking.

High levels of stress may make it harder to maintain self-control, especially when trying to control our unhealthy behaviors. Training on improving self control and decreasing stress may help decrease unhealthy behaviors. The goal of this new training program will be to decrease a subject's unhealthy behavior by helping them better manage their stress and improve their self control over unhealthy habits.

DETAILED DESCRIPTION:
This study proposes to pilot a mindfulness based affect-regulation treatment approach to improve self-control and physiological and biochemical indicators of stress, as well as decrease unhealthy/maladaptive behaviors such as drinking, overeating, and smoking. The broad aims of the treatment approach will be to teach participants to (1) observe and increase awareness of cognitive, affective, bodily sensations/expressions and action-urge components of emotional/compulsion experiences; and (2) develop alternate affective, behavioral and cognitive coping strategies in managing and regulating affect/urge experiences. It is hoped that the findings from this study will aid in the further development of treatment and prevention programs targeting stress reduction and coping to improve control over maladaptive behaviors and decrease physical and mental health symptoms.

Aims:

1. Develop a mindfulness based affect-regulation therapy manual, and training materials to train therapists on a treatment approach aimed at improving self-control over unhealthy addictive behaviors.
2. Develop and implement "Stress in Control" (SynC) training competence and adherence rating scales;
3. Conduct a preliminary study using the SynC manual, which will evaluate the effectiveness and feasibility of SynC in comparison to a Primary Care Treatment Control Group and a Historical Control Group approach for 100 individuals interested in help in decreasing targeted unhealthy behaviors. Primary outcomes will be a reduction in unhealthy problem behaviors, and secondary outcomes will be decrease in measures of stress, and increases in emotion regulation and self control.
4. (secondary aim) Collect baseline data on measures of self control, mood, coping, personality, cognitive functioning, acute and chronic stress, and mental and physical health on a large sample of subjects seeking help in decreasing unhealthy behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages 18-60 years;
2. Able to read and write;
3. Interested in treatment aimed at gaining greater control over an unhealthy, maladaptive behavior

Exclusion Criteria:

1. Any psychotic disorder or current psychiatric symptoms requiring specific attention, including active symptoms of psychosis or suicidal/homicidal ideation
2. Pregnant women will be excluded.
3. Inability to give informed consent
4. Traumatic brain injury or loss of consciousness
5. Medical problems requiring immediate attention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Development of treatment approaches | 1 year
  Develop a mindfulness based affect-regulation therapy manual, and training materials to train therapists on a treatment approach aimed at improving self-control over unhealthy addictive behaviors.
Measure effectiveness of intervention | 2 years
  Conduct a preliminary study using the SynC manual, which will evaluate the effectiveness and feasibility of SynC in comparison to a Primary Care Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States